CLINICAL TRIAL: NCT05592353
Title: Effect of Post-operative Brace on Pain and Patient Outcomes Following Hip Arthroscopy for FAIS: A Randomized Study
Brief Title: Effect of Post-operative Brace on Pain and Patient Outcomes Following Hip Arthroscopy for FAIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Weber (Other)
Responsible Party: Sponsor-Investigator, Alexander Weber, Assistant Professor, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-20-00060
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hip Arthroscopy
MeSH Terms: interventions — Braces

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brace (Active Comparator)
  Interventions: Other: Brace
- No Brace (No Intervention)

INTERVENTIONS:
Other: Brace — Brace following hip arthroscopy
  Arms: Brace

SUMMARY:
The routine application of hip brace following hip arthroscopy for femoroacetabular impingement syndrome (FAIS) has no proven clinical benefits. This study will investigate whether the application of hip brace affects the post-operative course and patient reported outcomes in patients undergoing hip arthroscopy for FAIS.

ELIGIBILITY:
Inclusion Criteria:

* Patient age of 18 years or older
* Patients with femoroacetabular impingement syndrome (FAIS) and who are candidates for surgical treatment with hip arthroscopy

Exclusion Criteria:

* Patient age < 18 years
* Patients with FAIS who are not surgical candidates (surgical therapy is not indicated)
* Patients with previous, ipsilateral hip procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hip Outcome Score | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Keck School of Medicine of the University of Southern California, Los Angeles, California, United States